CLINICAL TRIAL: NCT01220011
Title: A Cluster Randomized Trial Comparing a Conservative Management and Primary Laser Surgery
Brief Title: Randomized Controlled Trial Comparing a Conservative Management and Laser Surgery
Acronym: TTTS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K090601; ID RCB : 2010-A00026-33 (Other: AFSSAPS)
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Blood and Blood Disorders; Anemia, Neonatal; Hematologic Disease; Infant, Newborn, Diseases
Keywords: Fetoscopic Laser surgery; Stage 1 Twin - twin transfusion syndrome
MeSH Terms: conditions — Hematologic Diseases; Anemia, Neonatal; Infant, Newborn, Diseases; Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NO INTERVENTION (Experimental)
  Interventions: Procedure: Fetoscopic laser surgery
- fetoscopic laser (Active Comparator)
  Interventions: Procedure: Fetoscopic laser surgery

INTERVENTIONS:
Procedure: Fetoscopic laser surgery — Fetoscopic laser surgery

SUMMARY:
The objective of this trial is to compare both strategies (Expectative Vs Fetoscopic laser surgery) for patients with stage 1 TTTS and favorable obstetrical parameters in an international randomized controlled trial. This trial will answer an important question and will help in the management and tailoring of surgical indications in stage 1 TTTS.

DETAILED DESCRIPTION:
Although we demonstrated the overall benefit of fetoscopic laser surgery as first-line treatment in twin-twin transfusion syndrome (TTTS), indications in early stage TTTS are controversial. Indeed, a conservative management with close follow-up is offered in some centers as first-line management for QUINTERO stage 1 TTTS, although this strategy has not been formally compared to first-line fetoscopic placental surgery. The objective of this trial is to compare both strategies for patients with stage 1 TTTS and favorable obstetrical parameters in an international randomized controlled trial. Patients randomized to a conservative management will be followed on a weekly basis as long as the syndrome remains stable using obstetrical and fetal parameters and until an adequate gestational age is reached allowing delivery. Cases progressing to stage ≥ 2 or with a worsening of obstetrical parameters during follow-up in this group will be actively treated by percutaneous laser coagulation. Patients allocated to the "immediate laser" group will be treated by fetoscopic laser surgery within 24 h following randomization. The primary end-point encompasses survival and neurological morbidity at the age of 6 months for each foetus randomized. Analyses and power computations use a cluster-trial methodology that accounts for the inter-twin correlation, with many benefits over more traditional designs using a per-pregnancy outcome. With proportions of 60% and 75% meaning a clinically relevant difference of 15% between the groups, 200 fetuses or equivalently 100 pregnancies would be needed in each arm to reach a power of 80% with an alpha-risk of 5%, allowing 2 interim analyses based upon LAN-DEMETS boundaries and an O'Brien-Fleming function. Inclusion criteria, interventions and randomisation were investigated through a preliminary survey across potential participating centers. Based on this survey, it is anticipated that 3 years will be needed to achieve the requested number of patients. This trial will answer an important question and will help in the management and tailoring of surgical indications in stage 1 TTTS.

ELIGIBILITY:
Inclusion Criteria:

* TTTS stage 1 (Euro foetus criteria)
* Gestational age > 16 and < 26 weeks
* Age > 18
* Informed consent

Exclusion Criteria:

* Therapeutic amniocentesis prior to referral
* Short cervix < 15 mm on transvaginal US
* Severe maternal discomfort:Dyspnea and orthopnea, Abdominal pain > 4 on a 10-level visual analogic pain scale, Contractions > 1 per hour
* PPROM
* Fetal malformations unrelated to TTTS
* Follow-up is impossible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2011-04-19 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
survival and neurological morbidity at the age of 6 months for each foetus randomized | 6 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Yves VILLE, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (11):
- United States (8):
  - Children's Hospital Colorado and Colorado Fetal Care Center, Aurora, Colorado
  - University of MD /Department of Obstetrics, Gynecology & Reproductive Sciences, Baltimore, Maryland
  - Fetal Care Center of Cincinnati, Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Ohio State University / OSU Fetal Therapy Program, Columbus, Ohio
  - Fetal Diagnosis and Treatment, The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Fetal Treatment Program of New England, Hasbro Children's Hospital, The Warren Alpert Medical School of Brown University., Providence, Rhode Island
  - The Texas Fetal Center, Children's Memorial Hermann Hospital, University of Texas Medical School, Houston, Texas
  - Fetal Therapy Program, Evergrenn Hospital Medical Center, Kirkland, Washington
- Canada (2):
  - Mount Sinai Hospital, University of Toronto, Toronto, Ontario
  - Hospital Ste-Justine, Montreal, Quebec
- Necker Enfants Malades, Paris, France

REFERENCES:
- [Derived] Stirnemann J, Slaghekke F, Khalek N, Winer N, Johnson A, Lewi L, Massoud M, Bussieres L, Aegerter P, Hecher K, Senat MV, Ville Y. Intrauterine fetoscopic laser surgery versus expectant management in stage 1 twin-to-twin transfusion syndrome: an international randomized trial. Am J Obstet Gynecol. 2021 May;224(5):528.e1-528.e12. doi: 10.1016/j.ajog.2020.11.031. Epub 2020 Nov 26. PMID 33248135